CLINICAL TRIAL: NCT00594061
Title: Iowa/Nucleus 10/10 mm and Nucleus Freedom Cochlear Implants Implanted Bilaterally in Children Ages 12-24 Months
Brief Title: Iowa/Nucleus 10/10 mm and Nucleus Freedom Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruce J Gantz (Other)
Responsible Party: Sponsor-Investigator, Bruce J Gantz, Department Head --Department of Otolaryngology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200710716
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Results first posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss, Bilateral
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Bilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): There is no arm to this study--(each participant serves ashis or her own control). Blinding or masking procedures are not included in the design, as it is not possible to conceal the presence or absence of a cochlear implant from device recipients and/or clinical investigators.
  Interventions: Device: Iowa/Nucleus 10/10 mm and Freedom Cochlear Implantation

INTERVENTIONS:
Device: Iowa/Nucleus 10/10 mm and Freedom Cochlear Implantation — Participants will receive one standard Nucleus Freedom electrode array and an Iowa/Nucleus 10/10 mm electrode array on the contralateral side.

SUMMARY:
The purpose of this study is to evaluate whether the Iowa/Nucleus 10/10 mm in one ear, in conjunction with a Nucleus Freedom implant in the other ear can provide useful binaural hearing in pediatric subjects who have bilateral severe to profound hearing loss and meet the criteria for cochlear implantation. The Iowa/Nucleus 10/10 mm cochlear implant has a short, 10 mm electrode array that it is inserted only into the more basal region of the cochlea. Unlike a conventional cochlear implant, the Iowa/Nucleus 10/10 mm is expected to preserve the regions of the cochlear partition that are apical to the electrode, thus leaving them available for possible future advances in the field of otolaryngology and hearing devices, such as mammalian hair cell regeneration techniques or improved implantable hearing devices. The Iowa/Nucleus 10/10 mm will be implanted in the contralateral ear from the Nucleus Freedom electrode array as a means of providing bilateral stimulation of auditory pathways while preserving the middle and apical regions of the scala media.

DETAILED DESCRIPTION:
The study will be conducted as a repeated-measure , single-subject experiment. A single- subject research design (in which each participant serves as his or her own control) is appropriate because it accommodates the heterogeneity that characterizes hearing- impaired population s. Blinding or masking procedures are not included in the design, as it is not possible to conceal the presence or absence of a cochlear implant from device recipients and/or clinical investigators.

Preoperatively , candidates will be assessed with their current amplification to evaluate their appropriateness for entrance into the study. The candidates' audiometric configuration must meet the above inclusion criteria. That is, the candidate must have a severe-to-profound sensorineural hearing loss from 250 to 8000 Hz. Prior to testing, the appropriateness of the hearing aid fitting will be assessed and adjustments made if necessary. In cases where amplification has not been used for more than one year, new hearing aids will be fit, worn for a minimum three-month trial and the participants re- evaluated to confirm continuance with the study.

Participants will receive one standard Nucleus Freedom electrode array and an Iowa/Nucleus 10/ 10 mm electrode array on the contralateral side. Half will be implanted with the 10 mm electrode array on their right side and half will be implanted with the 10 mm electrode array on their left side. We will alternate every other subject between the right and left ears. Postoperatively, Iowa/Nucleus 10110 mm electrode alone, standard Freedom electrode alone, and bilateral listening (i.e., Iowa/Nucleus 10/ 10 mm and standard electrodes together) modes will be compared with repeated testing through five years of age of the child. These comparisons will help to evaluate the effects of bilateral stimulation using different cochlear implant devices while possibly preserving the scala media, organ of Corti, and supporting cells for future advances in the ear receiving the Iowa/Nucleus 10/ 10 mm electrode device. In addition, we will attempt to compare these results with age-matched unilaterally implanted children tested on the same speech perception and speech/language measures. In addition, if possible, we will attempt to compare speech perception and speech/language measures on age-matched children with bilateral standard long electrode arrays in both ears. The following defines the various modes referenced throughout the course of this text:

Iowa/Nucleus 10/10 mm Electrode Array: The Iowa/Nucleus 10/ 10 mm electrode array was designed to reduce the incidence of intracochlear injury and developed by the Iowa Cochlear Implant Team and Cochlear Americas. This array was designed to preserve the scala media, organ of Corti and supporting cells of the implanted ear for future advances in molecular and/or genetic treatments of the inner ear. This investigational device is very

similar to the Nucleus Hybrid-6 (formerly known as CI24RE Hybrid), the subject ofIDE No. 0990155. See ATTACHMENT 1 for a letter from the Sponsor ofIDE No. 0990155 authorizing the FDA to review the information in IDE No. 0990155 for purposes of the current IDE application. Like the Hybrid-6, the Iowa/Nucleus 10/ 10 mm cochlear implant is 0.2 mm x 0.4 mm in diameter and has a short, 10 mm electrode array that it is inserted only into the more basal region of the cochlea. In comparison to the Hybrid-6, the Iowa/Nucleus 10/ 10 mm cochlear implant has a total of 10 contacts, or 4 more than the 6 contacts/channels present on the Hybrid-6. The contacts are spaced closer together and occupy approximately 6 mm of the apical segment of the 10 mm array.

Nucleus Freedom electrode array: The standard electrode array, which is 19 mm in length.

Bilateral Stimulation :The use of the Iowa/Nucleus 10110 mm cochlear implant and the Nucleus Freedom cochlear implant on contralateral ears.

1.4 Preoperative Procedures: 1.4.1 Informed Consent: A preoperative interview will be conducted by the surgeon and audiologist to inform the parent(s) or legal guardian of the child about all aspects of implantation with the Iowa/Nucleus 10/10 mm cochlear implant and Nucleus Freedom cochlear implant, study expectations, number of visits, surgical procedure, as well as the postoperative evaluation schedule. The risks of surgery shall be explained to the parent(s) or guardian as outlined on the Informed Consent Form (Parental Agreement). These include the normal risks associated with general anesthetic, as well as other risks such as facial paralysis, dizziness, meningitis, postoperative discomfort, and flap complications. The potential limitations and advantages of implantation with the Iowa/Nucleus 10/10 mm and Nucleus Freedom cochlear implants shall also be explained. The parent(s) or guardian will be given adequate time to review the Informed Consent Form and given the opportunity to ask questions about the Informed Consent and/or the study prior to signing the Informed Consent Form. The parent(s) or guardian will then be given a copy of the signed Informed Consent Form.

Note that the Informed Consent Form must be reviewed and signed by the relevant parties prior to any study evaluation taking place. Any testing,for screening purposes, completed prior to consent being obtained must be repeated after theparticipant consents toparticipation in the study.

1.4.2 Hearing History: Information regarding P.articipant' s hearing-history (etiology, onset of hearing loss, duration of severe-to-profound hearing loss, amplification use) is to be reported.

1.4.3 Medical/Surgical History: The participant's medical/surgical history is to be reported and is required in order to determine that the participant is medically suitable for cochlear implantation .

Information to be collected may include: the participant 's general medical history, medications, radiological information (i.e. x-rays), otologic history, and otologic surgical history.

1.4.4 Fitting of Hearing Aids: Lack of benefit from appropriately fit hearing aids will be determined by the lack of progress in the development of simple auditory skills as defined by aided and unaided behavioral thresholds; auditory brainstem response testing; otoacoustic emission testing; steady state evoked potential testing; IT-MAIS and/or the lack of developmentally appropriate vocal behaviors. Criteria for appropriate vocal behaviors include achieving the production of canonical babble as defined by production of reduplicated sequences such as [mamama], [dadadal, or [bababal] (Oller and Eilers 1988). Hearing aid use will be determined by parental and educator reports.

Bilateral behind-the-ear (BTE) hearing aids will be used during the three month trial period. Audiometric criteria must be met with the participants using appropriately fit hearing aids. Ifthe participant has not been appropriately fit with amplification, hearing aids will be fit prior to the completion of aided audiometric testing to ensure that candidacy criteria are met.

The National Acoustics Laboratories' (NAL) and Desired Sensation Level (DSL), hearing aid fitting strategies will be used, depending upon the age of the candidate (Dillon, 1999; Scollie, et al, 2005) to assess the degree to which real-ear or coupler- predicted targets are met for each patient. These fitting methods are based on extensive research and clinical trials with patients with sensorineural hearing loss and are the most widely used fitting formulas in clinical use.

Real-ear measures or DSL measures will be made to verify that the target of the frequency response is within 5 dB per octave of the target measure.

For those candidates that wear hearing aids fit based on DSL targets, coupler-predicted maximum output levels at 90 dB HL will not be exceeded.

1.4.5 Audiological Assessment The degree of hearing loss will be determined by a combination of electrophysiological and behavioral tests including auditory brainstem response testing; otoacoustic emission testing; steady state evoked potential testing; behavioral observation audiometry, visual reinforcement audiometry and/or conditioned play audiometry. Audiological assessment will include unaided and aided audiometric thresholds.

Unaided audiometric thresholds will be obtained for each ear, using insert earphones when possible. Thresholds will also be obtained using the standard audiometric technique conditioned play audiometric (CPA) techniques, visual reinforcement audiometric (VRA) and/or behavioral observation (BOA) techniques for pure-tone air-conduction. The most appropriate testing technique will be used according to the child's age. Bone conduction testing will be completed using the above techniques. Aided audiometric thresholds will be obtained, using narrowband noise, for each ear in the sound-field using standard audiometric techniques, CPA, VRA or BOA with the speakers positioned at 45°-azimuth relative to the participant's head. Results for unaided testing must be reported for the frequencies of 250, 500, 1000, 2000, 4000, 6000, and 8000 Hz. Results for aided testing needs to be reported for the frequencies of 250, 500, 1000, 2000 and 4000 Hz.

A candidate is not considered enrolled until a properly executed Informed Consent form has been obtained and along with the results of the preoperative candidacy evaluation and reviewed and approved by the University of Iowa.

1.4.6 Baseline Speech Perception and Speech/Language Testing

In order to establish a baseline level of auditory function, auditory function will be evaluated in the best aided condition using the following battery of speech language production and subjective measures:

* The Infant-Toddler Meaningful Auditory Integration Scale (IT-MAIS) is a parent questionnaire that consists of ten questions regarding a young infant or toddler's auditory behavior , e.g. "Does the child spontaneously respond to his/her name in quiet with auditory cues?" Each question is scored on a five point scale: O=never, 1=rarely, 2=occasionally, 3=frequently, and 4=always . The aim of this tool is to assess the benefit of the child's personal amplification device(s). This questionnaire is generally used during the cochlear implant work-up to assess hearing aid benefit. It is also used post-cochlear implantation to chart the progress the child is making with his/her cochlear implant when other formalized speech perception tests are not appropriate.
* Vocalizations/speech sample protocol: The samples will be elicited by presenting the child with a set of age-appropriate toys with lexical labels that have phonemes representing early consonant productions and the entire vowel quadrilateral. Additionally, for children who are beginning to combine consonant and vowel productions and likely to be between 18 and 29 months of age, we will use the assessment words included in previous research conducted by Preisser, Hodson and Paden (1988). This word list assesses 20 consonants, and all classes of phonemes, plus 10 consonant clusters. The words will be elicited by objects or questions. Elicited productions will be transcribed using broad International Phonetic Alphabet transcription. A number of analyses will be completed in order to describe the patterns of speech acquisition. We will use independent analyses (Stoel-Gammon & Dunn, 1985), allowing us to describe the sounds and syllable structures produced by each child.

Specifically, we will analyze each participant's phonemic inventory in the initial and final position with respect to place and manner of production rather than phonemic target. We will also use relational analyses, from the point at which we obtain 90 different words. We will then compare the child's production with the standard adult phonemic target. Speech development will be assessed using the Percent Phoneme Correct and Percent Vowel Correct (PPC or PVC ) {Shriberg and Kwiatkowski, 1982). When developmentally appropriate, phoneme production skills will also be assessed using the Goldman-Fristoe Test o(Articulation-2 (Goldman & Fristoe, 2000). This measure has norms based on the performance of normal-hearing children from age 2 years to 21 years.

* MacArthur Communicative Developmental Inventories (CD!) and the Minnesota Child Development Inventor y (MinnCDI, Ireton & Thwing, 1974) are parent report measures that provide an index of growth from birth to 30 months of age. The CD!has a ceiling on the Wordsand Sentences version of 30 months of age; however the MinnCDI assesses development up to 6 years of age. The CD!also has two forms: Gestures and Words for children aged 8- to

  16-months-old and Words and Sentences for children aged 17- to 30-months- old. In order to create a single scale for these two measures, an item analysis using item response theory (Drasgow, & Parsons, 1983) will be performed and the scores will be transformed to a Rasch ability scale that provides a single equal-ability-interval scale suitable for growth curve analysis.
* The Preschool Languag e Scale-3 (PLS-3) (Zimmerman, Steiner, & Pond 1992) is a standardized language test that is used to measure the language development of children with normal hearing aged 0 months to 83 months. The test evaluates "Expressive Communication" and "Auditory Comprehension" and is designed to evaluate skills in a variety of areas: vocal development, social communication , attention, semantics (content), structure (form), and integrative thinking skills.

1.4.7 Surgical Procedure: The surgical procedure for the Iowa/Nucleus 10/ 10 mm cochlear implant is different from the Nucleus Freedom cochlear implant. The surgical procedure for the Iowa/Nucleus l 0/10 mm requires care to prevent inner ear damage. The cochleostomy is smaller (approximately 0.5 mm in diameter compares to > 1.0 mm for the Nucleus Freedom electrode). Soft surgery techniques will be used on both. The cochleostomy will be made in a similar position for both devices. Creation of the cochleostomy requires control of bleeding and removal of bone over the scala tympany exposing the endosteum. The endosteum is removed with a .02 mm hook. No suctioning of perilymph is allowed. The devices are then advanced slowly into the cochlea. For the Iowa/Nucleus 10/ 10 mm cochlear implant, the array is inserted 10 mm into the scala tympani and 19 mm for the Nucleus Freedom cochlear implant. Intraoperative impedance telemetry measurements will beperformed using CG,MPJ , MP2 and MP1+2 modes. The postoperative hospital stay is usually <23 hours.

1.5 Postoperative Procedures: 1.5.1 Device Activation The participants will be fit with Freedom speech processors using a behind-the-ear (BTE) controller or body level controller. Speech processing strategies used with this device will include ACE (RE), ACE, CIS (RE), CIS or SPEAK, which are all FDA approved for children . Threshold (T) and comfort (C) values will be measured for the electrical stimulation for each of the channels (10 on the Iowa/Nucleus 10/ 10 mm and 24 on the Nucleus Freedom). Impedance telemetry results using common ground (CG) and monopolar (MPI , MP2 and MP 1+2) stimulation modes will also be recorded . This information will be used to program the speech processor and also to monitor the device for possible degradation of function and/or damage to neural elements.

The process of adjusting the speech processor programs takes place over a period of several months for young children. Techniques used for programming speech processors of young children are standard audiological techniques for children in this age group and require two audiologists to perform . Play audiometry techniques will be used, as appropriate for the child's developmental level, to determine electrical threshold levels for the channels in a child's program. Behavioral observation or visual reinforcement

audiometry will be used for children who are unable to perform play audiometry. Electrophysiological data will verify levels obtained behaviorally or in those instances when behavioral information is limited. Electrical comfort levels will be set conservatively on initial programs to ensure a comfortable listening level for the child. Levels will be increased gradually at home and over several programming sessions during the first year of implant use. This approach is necessary in order to ensure comfortable listening levels are not exceeded in children who are unable to give us direct input as to how loud sounds are through the cochlear implant.

Parents and professionals working with the children will receive extensive counseling regarding how the equipment functions, maintenance and troubleshooting of the device, and progression of auditory skills of children who cochlear implants. This is accomplished during visits to the center and through in-service training offered locally via the fiberoptic teleconferences.

1.5.2 Programming Follow-up Following surgical implantation of the device and an adequate healing period, the implants will be activated (usually 4 to 6 weeks after surgery) and programmed. Thereafter, prior to the 4-month post-operative evaluation, three additional programming follow-up sessions will be scheduled at 2 weeks, 1 month, and 2 months as it is not unusual for threshold and comfort levels to change during the initial postactivation period. The follow-up sessions will allow the participant 's T- and C-levels to be checked as well as any programming adjustments to be made based on the participant's initial experience with the device. Electrical impedance measures also will be obtained.

Additional programming at additional postactivation intervals will be assessed and conducted as needed.

1.5.3 Listening conditions

The following describes the listening modes used by the child during each speech perception or speech/language measure:

* Iowa/Nucleus 10/10 mm electrode array only (unilateral),
* Nucleus Freedom electrode array only (unilateral),
* Iowa/Nucleus 10/ 10 mm and Nucleus Freedom electrodes together (bilateral).

1.5.4 Speech Perception and Speech/Language Testing: Speech perception and speech/language development will be assessed longitudinally at 4, 8, 12, 18, 24 months, and annually thereafter through five years of age. The tests or questionnaires will be administered age appropriately.

1.5.4.1 Speech Perception

* The Infant-Toddler Meaningful Auditor y Integration Scale {!T-MAIS) or Meaningful Auditory Integration Scale (MAIS) is a parent questionnaire that consists of ten questions regarding a young infant or toddler's auditory behavior, e.g. "Does the child spontaneously respond to his/her name in quiet with auditory cues?" Each question is scored on a five point scale: O=never,

  1. rarely , 2=occasionally, 3=frequently, and 4=always. The aim of this tool is to

     assess the benefit of the child's personal amplification device(s). This questionnaire is generally used during the cochlear implant work-up to assess hearing aid benefit. It is also used post-cochlear implantation to chart the progress the child is making with his/her cochlear implant when other formalized speech perception tests are not appropriate.
* The Glendonald Auditor y Screening Procedure Word Test (GASP) contains 12 single-syllable and multisyllable words. The child will be tested in the bilateral listening condition. This test is always administered in a live-voice mode. The child is asked to repeat the word presented by the clinician. The child is encouraged to use sign if his or her verbal approximations are not clear to the clinician. This test is the easiest open-set measure in this battery because it includes common vocabulary and the speaker is familiar. It can be administered to children as young as two years of age.
* Iowa Children's Vowel Test requires the identification of a monosyllabic word from a closed set of four words (e.g., toe, toy, tie, two) varying only in vowel content (place and height). Ifthe child performs at 80% or higher, multi-talker babble at a +7 dB-C SIN will be added. It will be administered in both the unilateral and bilateral listening conditions at 70 dB C.
* The CID Four Choice Spondee and Monosyllable tests require the identification of a spondee or monosyllable from a set of four spondees (i.e., French fry, airplane, hotdog, popcorn) or monosyllables (i.e., ball, book, bird, boat), respectively presented in quiet. The CID test will be scored as total number of words correct. It will be administered in both the unilateral and bilateral listening conditions at 70 dB C.
* The CRISP JR. Test will be used to assess speech perception in noise in both the unilateral and bilateral listening conditions for children ages 2.5-5 years. This test is designed with 12 monosyllabic and 4 bi-syllabic words that are within the receptive language and vocabulary of 2.5- to 3.0-year-old children (Garadat & Litovsky, 2007). This test was developed and is licensed from the University of Wisconsin - Madison . Speech perception will be measured using a four- alternative forced choice paradigm. Target speech and background two-talker female babble will be presented from the front (0 degrees). Speech reception thresholds are measured adaptively using a three-down/one-up algorithm finding the 79.4% correct level.
* The Multisyllabic Lexical Neighborhood Test (MLNT) and Lexical Neighborhood Test (LNT) are two open-set word recognition tests. The experimenter gives a list of 24 words and the participants are expected to repeat the word after each presentation. The MLNT consists of two parallel lists. The LNT and MLNT are based on the lexical characteristics of word frequency and neighborhood density, and include words found in the vocabularies of children age three to five.

1.5.4.2 Speech and Language Testing -all administered in the bilateral listening condition

* Vocalizations/speech samples as described above in baseline/pre-operative testing will be collected.
* MacArthur Communicative Developmental Inventories (CDI) and the Minnesota Child Development Inventory (MinnCDI, Ireton & Thwing, 1974) as described above in baseline/pre-operative testing will be collected.
* The Preschool Language Scale-3 (PLS-3), Zimmerman, Steiner, & Pond, 1992) as described above in baseline/pre-operative testing will be collected.
* The child's mean length of utterance (MLU) and number of different words (NDW) will be computed a speech sample of at least 50 utterances and will be based upon 100 utterances once this level of production is reached.
* Peabod y Picture Vocabulary Development Scale. This is a receptive vocabulary test that will be administered in an auditory/visual condition. The test provides an index of receptive vocabulary skill.
* Ex pressive Vocabulary Test. This is an expressive vocabulary test that provides an index of expressive vocabulary skill.

1.5.5 Psychophysical and Electrical Impedance Measurements: The following psychophysical and electrical impedance measurements will be attempted at 4, 8, 12, 18, 24 months, and annually there after through five years of age.

1. Electrical thresholds measured in current level.
2. Electrical maximum comfort levels measured in current level.
3. Impedance telemetry results using common ground (CG) and monopolar (MPI, MP2, MP I +2) stimulation modes.

Because this is a feasibility study, we will only be implanting up to 10 children. We recognize that this small number of subjects may not afford us enough statistical power to adequately answer all questions associated with using an Iowa/Nucleus 10/ 10 mm and a Nucleus Freedom electrode array in contralateral ears in pediatric subjects who have bilateral severe to profound hearing loss. However, it may lend us foundational knowledge to assess whether the Iowa/Nucleus 10/ 10 mm and Nucleus Freedom implants can provide useful bilateral hearing while at the same time preserving the scala media, organ of Corti and supporting cells of the ear implanted with the Iowa/Nucleus 1Oil0 mm array for future advances in molecular and/or genetic treatments of the inner ear.

ELIGIBILITY:
Inclusion Criteria:

* Twelve to twenty-four months of age at the time of implantation.
* Audiometric thresholds for frequencies 250 to 8000 Hz in the severe-to-profound hearing range bilaterally. The type of hearing loss must be categorized as sensorineural in nature.
* English spoken as a primary language (mono-lingual English speaking family, where English is the primary language).
* Willingness to comply with all study requirements.
* Multiple visits may be necessary preoperatively and/or postoperatively for data collection due to age and attention.
* Minimum of three month hearing aid trial.
* Patent cochlea and normal cochlear anatomy as shown by a CT Scan. It is standard clinical practice to perform a CT Scan on any patient pursuing cochlear implantation.
* Must be in a habilitation/educational program with an emphasis on spoken language development.

Exclusion Criteria:

* Medical or psychological conditions that contraindicate undergoing surgery.
* Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array.
* Developmental disabilities or other conditions that would prevent or restrict participation in the audiological evaluations and clinical trial.
* Hearing loss of neural or central origin.
* Unrealistic expectations on the part of the candidate and/or candidate's family,regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure(s) and prosthetic devices.
* Unwillingness or inability of the candidate to comply with all investigational requirements.
* Active middle ear infection.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2007-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J Gantz, MD, Principal Investigator — University of Iowa Department of Otolaryngology Pediatric Cochlear Implant Program
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Iowa/Nucleus 10/10 mm and Freedom Cochlear Implantation: There is no arm to this study--(each participant serves as his or her own control). Blinding or masking procedures are not included in the design, as it is not possible to conceal the presence or absence of a cochlear implant from device recipients and/or clinical investigators.
  Iowa/Nucleus 10/10 mm and Freedom Cochlear Implantation: Participants will receive one standard Nucleus Freedom electrode array and an Iowa/Nucleus 10/10 mm electrode array on the contralateral side.
Period: Overall Study
Arm/Group | Iowa/Nucleus 10/10 mm and Freedom Cochlear Implantation
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Iowa/Nucleus 10/10 mm and Freedom Cochlear Implantation: There is no arm to this study--(each participant serves ashis or her own control). Blinding or masking procedures are not included in the design, as it is not possible to conceal the presence or absence of a cochlear implant from device recipients and/or clinical investigators.
  Iowa/Nucleus 10/10 mm and Freedom Cochlear Implantation: Participants will receive one standard Nucleus Freedom electrode array and an Iowa/Nucleus 10/10 mm electrode array on the contralateral side.
Arm/Group | Iowa/Nucleus 10/10 mm and Freedom Cochlear Implantation
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9
Infant-Toddler Meaningful Auditory Integration Scale (IT-MAIS) [Mean (Standard Deviation); unit: units on a scale] — The IT-MAIS is a structured interview schedule used to assess the child's spontaneous responses to sound in his/her everyday environment. It consists of 10 questions with a total scale range of 0-40. Performance is scored in terms of the total number of points accrued out of 40 possible points. Higher score indicates better performance. Each question has a potential of 0 (lowest) to 4 (highest) points.
  units on a scale | 2.6 (5.5)
MacArthur Communicative Developmental Inventories (CDI) [Mean (Standard Deviation); unit: months] — The CDI is a parent report measure evaluating children's communicative development. The CDI Words and Gestures (WG) tests children aged 8- to 16-months. WG assesses the child's production of language by their responses to familiar words and phases. Raw scores are converted into age-equivalent scores.The maximum range of age equivalent scores is <8 months to 18 months. Higher age-equivalent scores indicate better outcomes.
  months | 10.4 (2.19)
Minnesota Child Development Inventory [Mean (Standard Deviation); unit: months] — This parent inventory consists of 54 statements describing the behaviors of infants and preschool-age children and provides measures of the child's expressive language development. The parent is asked yes/no questions and indicates whether the child is able to do what the statement says. Raw scores are converted into age-equivalent scores. The maximum range of age equivalent scores is 1 month to 63 months. Higher age-equivalent scores indicates better performance.
  months | 11.3 (2.6)
Preschool Language Scale-3 [Mean (Standard Deviation); unit: units on a scale] — Assesses global language skills using toys and pictures. This test assess auditory comprehension and expressive communication and a total language score is calculated. A higher total score indicates better performance. The standard score ranges from 50 to 150. A raw score for total language is calculated and converted into a standard score.
  units on a scale | 74.2 (8.1)

OUTCOME MEASURES:

1. Primary Outcome: Pre-school Language Test
Description: Assesses global language skills using toys and pictures. This test assess auditory comprehension and expressive communication and a total language score is calculated. The reported score was assessed at 48 months post-implantation. The total language standard score ranges from 50-150. A higher total score indicates better performance. A raw score for total language is calculated and converted into a standard score.
Time Frame: 48 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Iowa/Nucleus 10/10 mm and Freedom Cochlear Implantation
Number analyzed (Participants) | 8
units on a scale | 82.4 (22.7)

2. Secondary Outcome: Phonemically Balanced-Kindergarten Test (PB-K)-Bilateral
Description: PB-K Test was constructed to be an open-set test of word understanding for children. It is scored as a percentage of words correct. The test was measured using the Iowa/Nucleus 10/10 mm and Nucleus Freedom together, the Iowa/Nucleus 10/10 mm only, and the Nucleus Freedom electrode only conditions. The higher the score, the better the word understanding. The post-operative time point for this score was reported on average at 56 months post-implantation.
Time Frame: 56 months
Measure: Mean (Standard Error); unit: percentage of words correct
Arm/Group | Iowa/Nucleus 10/10 mm and Freedom Cochlear Implantation
Number analyzed (Participants) | 8
percentage of words correct
  bilateral | 85.7 (3.31)
  short electrode | 55.6 (7.9)
  long electrode | 85.9 (2.33)

ADVERSE EVENTS:
Time Frame: Following surgical implantation of the device and longitudinally at 4, 8, 12, 18, and 24 months, and annually thereafter through five years of age.
Arm/Group | Iowa/Nucleus 10/10 mm and Freedom Cochlear Implantation
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iowa/Nucleus 10/10 mm and Freedom Cochlear Implantation (N=9)
Failed device (Ear and labyrinth disorders) | 1 — Nine months post-implantation the child was seen in our clinic for swelling on his right cochlear implant site. The child underwent explantation of the device on his right side and was later re-implanted with a second Nucleus Freedom device.
Failed Device (Ear and labyrinth disorders) | 1 — Due to asymmetry in speech perception scores and electrical shorts with device, explantation of the device and reimplantation with a different device was recommended. Device failure report indicated a failed device due to electrode lead malfunction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No